CLINICAL TRIAL: NCT05454293
Title: One Talk at a Time: A Racial-ethnic Socialization Intervention for Diverse Families to Reduce Psychosocial Inequalities
Brief Title: One Talk at a Time: A Racial-ethnic Socialization Intervention for Diverse Families
Acronym: OTAAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Gabriela Stein, Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202064
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms; Anxiety Disorders and Symptoms; Behavioral Symptoms; Ethnic-Racial Socialization
Keywords: Ethnic-racial socialization; Race; Ethnicity; Discrimination; Diverse families; Cultural socialization; Preparation for bias; Culture; Parent-Child communication
MeSH Terms: conditions — Depression; Anxiety Disorders; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTAAT (Experimental): This group will receive the One Talk at a Time curriculum.
  Interventions: Other: One Talk at a Time: Race
- Parent-Child Communication (Active Comparator): This group will receive a curriculum focused on tips and strategies for navigating difficult topics with one's children such as current events and dating.
  Interventions: Other: One Talk at a Time: General

INTERVENTIONS:
Other: One Talk at a Time: Race — This intervention consists of short videos that include didactic modules and social modeling for having conversations with children about race, ethnicity, culture, and discrimination. The total intervention takes approximately 1.5-2 hours to complete online, and parents can move through the videos at their own pace.
  Arms: OTAAT
Other: One Talk at a Time: General — This intervention consists of short videos that include modules and handouts with tips for parent-child communication strategies for navigating difficult topics, such as dating and current events.
  Arms: Parent-Child Communication

SUMMARY:
This study is a randomized effectiveness trial that tests the online delivery of a video-based intervention (One Talk at a Time (OTAAT)) relative to a control group over a one-year span. Hypotheses include: 1.) The OTAAT intervention will increase parental motivation to engage in racial-ethnic socialization (RES) conversations, their skills and confidence in having these conversations, and the frequency and quality of these conservations; 2.) The OTAAT intervention will increase youth reports of their coping with discrimination, perceived efficacy in coping with discrimination in the future, ethnic-racial identity, and youth mental and academic outcomes; 3.) Greater parental discrimination and youth discrimination will moderate links between OTAAT intervention and parental ethnic-racial motivation + competency as well as youth ethnic-racial identity, coping, and psychosocial outcomes.

DETAILED DESCRIPTION:
This study will employ a mixed methods longitudinal randomized control trial design. All parents and youth will be assessed at four time points (Baseline, 3-month, 6-month, and 12-month) using surveys. Investigators will also use an observational racial-ethnic socialization (RES) task at 3-months to complement self-report data where parents and youth will have taped RES conversations.

Investiagtors will collect data with two balanced cohorts (Cohort 1 and Cohort 2). Parent-youth dyads (N=312) will be recruited through community-based organizations and diverse, public middle schools to reach a representative population of each racial-ethnic group. Specific recruitment procedures are included below.

Once an identified parent-youth dyad is recruited into the study, parents and youth will complete separate Qualtrics baseline surveys online. Parents will then receive either the intervention or the control materials via email or text within 2 weeks (and be given a month to start intervention). OTAAT consists of 11 videos (3-5 minutes each) that include didactic modules and social modeling. The total intervention takes approximately 1.5-2 hours to complete online, and parents can move through the videos at their own pace. The control condition will receive web-based communication materials onsite, including communication videos. Subsequent research follow-ups will occur at 3-months, 6-months, and 12-months with both parents and youth via Qualtrics.

After the initial intervention, parents will receive 6 additional OTAAT contacts via text messages/newsletters that will be spread out across the year with contacts at 1, 2, 4, 5, 8, and 10 months after the initial intervention. These contacts will include a short survey assessing the use of Ready, Set, Talk skills and setting times for having RES conversations. Parents in the control condition will similarly receive text messages/newsletters at the same time points.

At 3-month follow-up, parents and youth will also complete a video-recorded RES observational task via a virtual platform or in-person depending on family preference. During the observational task, parents and their children will be asked to spend five minutes discussing four discrimination encounters. During these conversations, parents will be asked to talk to their child about race and culture as they would at home in a natural manner. The task will take approximately 25-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child between the ages of 11 and 13
* Parental race/ethnicity either of East Asian, African American, Latinx (Central American) background
* Both parents are from the same pan-ethnic group

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Parental Motivation (Parent-reported) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  The study will use an adapted version of the Motivation to Change measure (Miller & Johnson, 2008) to assess parental motivation to engage in racial-ethnic socialization with their children.
Parental Skill (Parent-reported) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  The study will use the Racial Socialization Competency Scale (RaSCS; Anderson et al., 2019) to measure parental-perceived skill in delivering racial-ethnic socialization messages
Parental Confidence (Parent-reported) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  The study will use a recently developed scale (under review) that assesses how confident parents feel delivering racial-ethnic socialization messages
Coping with Discrimination (Youth-reported) Youth Coping with Discrimination | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's use of coping strategies will be measured using the Discrimination Coping Strategies Scale (Umaña-Taylor et al., 2008)

SECONDARY OUTCOMES:
Cultural Socialization Frequency (Parent and youth report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Frequency of cultural socialization messages will be measured using the cultural socialization subscale of the Ethnic-Racial Socialization Scale (Hughes & Chen, 1997). The measure will be adapted to measure frequency over the last 3 months rather than year.
Preparation for Bias Frequency (Parent and youth report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Frequency of preparation for bias messages will be measured using the preparation for bias subscale of the Ethnic-Racial Socialization Scale (Hughes & Chen, 1997). The measure will be adapted to measure frequency over the last 3 months rather than year.
Cultural Socialization Quality | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Quality of cultural socialization messages will be assessed during observational coding of parent-child discussions around scenarios describing experiences of discrimination. Coding will be based on Smith Bynum et al.'s (2016) scale.
Preparation for Bias Quality | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Quality of preparation for bias messages will be assessed during observational coding of parent-child discussions around scenarios describing experiences of discrimination. Coding will be based on Smith Bynum et al.'s (2016) scale.
Youth Self-Esteem (Youth and parent report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's self-esteem will be assessed using the Rosenberg (1979) measure
Youth Depressive symptoms (Youth and parent report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's current depressive symptoms will be measured using the PROMIS Pediatric Short-Form of Depressive Symptoms (Irwin et al., 2010)
Youth Anxiety symptoms (Youth and parent report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's current anxiety symptoms will be measured using the PROMIS Pediatric Short-Form of Anxiety Symptoms (Irwin et al., 2010)

OTHER OUTCOMES:
Youth Academic Motivation (Youth and parent report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's academic motivation will be measured using the Eccles (1983) scale
Youth Behavioral Symptoms (Youth and parent report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's behavioral symptoms will be assessed using the Misconduct Scale (Feldman et al, 2011)
Youth Racial-Ethnic Identity (Youth-report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's racial-ethnic identity will be assessed using the Multigroup Ethnic Identity Measure Sladeck et al., 2020)
Youth Racial-Ethnic Exploration (Youth-report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's racial-ethnic exploration will be assessed with the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015)
Youth Coping Efficacy (Youth-report) | Baseline, 3-month after intervention, 6-months after intervention, and 12-months after intervention
  Youth's coping efficacy will be measured using items developed for this study

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Livas Stein, PhD, Principal Investigator — University of Texas at Austin; Stephanie Coard, PhD, Principal Investigator — University of North Carolina, Greensboro; Lisa Kiang, PhD, Principal Investigator — Wake Forest University
Locations (1):
- University of North Carolina Greensboro, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No